CLINICAL TRIAL: NCT02339090
Title: Comparison of Somavaratan (VRS-317), a Long-acting Human Growth Hormone, to Daily rhGH in a Phase 3, Randomized, One-year, Open-label, Multi-center, Non-inferiority Trial in Pre-pubertal Children With Growth Hormone Deficiency
Brief Title: Long-Acting Growth Hormone in Children Compared to Daily rhGH
Acronym: VELOCITY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Versartis Inc. (Industry)
Responsible Party: Sponsor
Organization: Aravive, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14VR4
Record Dates: First submitted 2015-01-07; First posted 2015-01-15 (Estimated); Results first posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-11

CONDITIONS: Growth Disorders
Keywords: VRS-317; Growth Hormone Deficiency; Long Acting Recombinant Growth Hormone; Long Acting Growth Hormone; Pediatric Growth Hormone Deficiency; Growth Hormone Replacement Therapy; Versartis; Xten; Human Growth Hormone; somavaratan; growth failure
MeSH Terms: conditions — Growth Disorders; Dwarfism, Pituitary; Failure to Thrive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Somavaratan (Experimental): Participants will receive somavaratan 3.5 milligrams (mg)/kilogram (kg) subcutaneous (SC) bolus injection twice monthly for 12 months.
  Interventions: Drug: Somavaratan
- rhGH (Active Comparator): Participants will receive commercially available rhGH (genotropin) 34 micrograms (μg)/kg once daily SC bolus injection for 12 months.
  Interventions: Drug: rhGH

INTERVENTIONS:
Drug: Somavaratan — Somavaratan will be administered per dose and schedule specified in the arm description.
  Other Names: Long-acting recombinant human growth hormone; VRS-317
  Arms: Somavaratan
Drug: rhGH — rhGH will be administered per dose and schedule specified in the arm description.
  Other Names: daily growth hormone; recombinant growth hormone therapy
  Arms: rhGH

SUMMARY:
The trial will compare a twice-monthly somavaratan dosing regimen for non-inferiority of treatment effect against daily injections of rhGH.

DETAILED DESCRIPTION:
This study is designed as a pivotal study to compare the safety and efficacy of a selected dose regimen of somavaratan to daily rhGH. The study is a randomized, multi-center, open label study of 12 months duration. The primary endpoint is height velocity at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Chronological Age ≥ 3.0 years and ≤ 10.0 (girls) and ≤ 11.0 (boys).
* Pre-pubertal status: Absent breast development in girls, testicular volume < 4.0 mL in boys.
* Diagnosis of growth hormone deficiency (GHD) as documented by two or more growth hormone (GH) stimulation test results ≤ 10.0 ng/mL.
* Height standard deviation score (SDS) ≤ -2.0 at screening.
* Weight for Stature ≥ 10th percentile.
* Insulin-like growth factor-I (IGF-I) SDS ≤ -1.0 at screening.
* Delayed bone age (≥ 6 months).

Exclusion Criteria:

* Prior treatment with any growth promoting agent
* History of, or concurrent significant disease (for example, diabetes, cystic fibrosis, renal insufficiency).
* Chromosomal aneuploidy, significant gene mutations (other than those that cause GHD) or confirmed diagnosis of a named syndrome.
* A diagnosis of Attention Deficit Hyperactivity Disorder.
* Daily use of anti-inflammatory doses of glucocorticoid.
* Prior history of leukemia, lymphoma, sarcoma or cancer.
* Treatment with an investigational drug in the 30 days prior to screening.
* Known allergy to constituents of the study drug formulation.
* Ocular findings suggestive of increased intracranial pressure and/or retinopathy at screening.
* Significant spinal abnormalities including scoliosis, kyphosis and spina bifida variants.
* Significant abnormality in screening laboratory studies

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 138 (Actual)
Dates: Start 2015-08-26 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2017-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Will Charlton, MD, Study Director — Sponsor GmbH

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were stratified by region (North America and Europe), age (above and below anticipated median age of 7.5 years) and baseline Insulin-like growth factor-I (IGF-I) standard deviation score (SDS) (above and below anticipated median of -1.7) and randomized in a 3:1 ratio to receive either somavaratan or recombinant human growth hormone (rhGH).
Groups:
- Somavaratan: Participants received somavaratan 3.5 milligrams (mg)/kilogram (kg) subcutaneous (SC) bolus injection twice monthly for 12 months.
- rhGH: Participants received commercially available rhGH (genotropin) 34 micrograms (μg)/kg once daily SC bolus injection for 12 months.
Period: Overall Study
Arm/Group | Somavaratan | rhGH
Started | 104 | 34
Received a Least 1 Dose of Study Drug | 104 | 32
Completed | 98 | 29
Not Completed | 6 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Non-compliance With Study Drug | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Poor Growth | 3 | 0
Not completed — Randomized but not treated | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received any amount of study drug.
Groups:
- Somavaratan: Participants received somavaratan 3.5 mg/kg SC bolus injection twice monthly for 12 months.
- rhGH: Participants received commercially available rhGH (genotropin) 34 μg/kg once daily SC bolus injection for 12 months.
- Total: Total of all reporting groups
Arm/Group | Somavaratan | rhGH | Total
Number analyzed (Participants) | 104 | 32 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.0 (2.03) | 6.9 (2.38) | 7.0 (2.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 10 | 56
  Male | 58 | 22 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 3 | 11
  Not Hispanic or Latino | 96 | 29 | 125
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 5 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 91 | 31 | 122
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Annual Height Velocity
Description: Height measured without shoes in triplicate by stadiometer. Annual height velocity was calculated as (height at Month 12 - height at Baseline)/(Month 12 Date - Baseline Date) * 365.25, where height was expressed as centimeters (cm) so that height velocity is expressed as centimeters per year (cm/yr). Annual height velocity after 12 months continuous treatment with either somavaratan or daily rhGH has been reported. Missing data was imputed using last observation carried forward. Least square (LS) mean was calculated using analysis of covariance (ANCOVA) model.
Time Frame: 12 months
Population: ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: cm/year
Arm/Group | Somavaratan | rhGH
Number analyzed (Participants) | 104 | 34
cm/year | 9.43 (0.28) | 10.70 (0.48)
Statistical Analysis 1: Comparison: Somavaratan vs rhGH; An ANCOVA model will be used to determine the adjusted (least squares) means and standard error (SE) to determine the confidence interval (CI) of the difference. ANCOVA model included treatment group, region, and gender as fixed effects; with baseline age and baseline IGF-I SDS as covariates; Test type: Non-Inferiority — Threshold for significance: annualized height velocity between somavaratan and daily rhGH ≤ -2.0 cm/year; LS Mean Difference = -1.28, 95% CI 2-sided [-2.32 to -0.24]

2. Secondary Outcome: Change From Baseline in Height Standard Deviation Score (SDS) at Month 12
Description: Height SDS was determined using the Center for Disease Control (CDC) Clinical Growth Charts; 2000. The SD score was calculated as the participant's height value minus the mean divided by the standard deviation (SD). The mean and the SD vary depending on the age and sex of the participant. Mean change from baseline in height SDS at Month 12 is presented.
Time Frame: Baseline, Month 12
Population: ITT population included all randomized participants. Here, 'overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Somavaratan | rhGH
Number analyzed (Participants) | 98 | 30
SD score | 0.8 (0.53) | 1.0 (0.51)

3. Secondary Outcome: Change From Baseline in Bone Age Relative to Chronological Age at Month 12, as Assessed by Central Reader
Description: Bone age was assessed from a radiograph of the left hand and wrist by central reader.
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Somavaratan | rhGH
Number analyzed (Participants) | 98 | 29
months | 1.1 (0.47) | 1.3 (0.55)

4. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) at Month 12
Description: The BMI is a person's weight in kilograms (kg) divided by the square of height in meters.
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Somavaratan | rhGH
Number analyzed (Participants) | 99 | 30
kg/m^2 | 1.1 (0.86) | -0.1 (0.95)

5. Secondary Outcome: Change From Baseline in Body Weight at Month 12
Description: Body weight measured in light clothing and without shoes.
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Somavaratan | rhGH
Number analyzed (Participants) | 100 | 30
kg | 4.9 (1.87) | 3.8 (1.64)

6. Secondary Outcome: Change From Baseline in Insulin-like Growth Factor 1 (IGF-I) SDS at Month 12
Description: The SD score was calculated as the actual value of IGF-I minus mean reference value of IGF-1 divided by reference standard deviation of IGF-I. The mean and the SD vary depending on the age and sex of the participant. Change in IGF-I level (SD score) at Month 12 from Baseline was assessed. A higher score reflects a better outcome.
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Somavaratan | rhGH
Number analyzed (Participants) | 98 | 28
SD score | 0.9 (0.99) | 1.8 (0.72)

7. Secondary Outcome: Change From Baseline in Insulin-like Growth Factor Binding Protein 3 (IGFBP-3) at Month 12
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: nanomoles (nmol)/milliliter (mL)
Arm/Group | Somavaratan | rhGH
Number analyzed (Participants) | 90 | 26
nanomoles (nmol)/milliliter (mL) | 32.2 (30.2) | 49.8 (19.1)

8. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. SAEs included death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of serious and non-serious AEs regardless of causality is located in 'Reported Adverse Events module'.
Time Frame: Baseline up to Month 12
Population: Safety population included all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Somavaratan | rhGH
Number analyzed (Participants) | 104 | 32
Participants | 80 | 22

ADVERSE EVENTS:
Time Frame: Baseline up to Month 12
Description: Safety population included all participants who received any amount of study drug.
Arm/Group | Somavaratan | rhGH
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/32
Serious Adverse Events (participants affected / at risk) | 6/104 | 0/32
Other Adverse Events (participants affected / at risk) | 59/104 | 16/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Somavaratan (N=104) | rhGH (N=32)
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 2 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Syringomyelia (Nervous system disorders) | 1 | 0
Glomerulonephritis (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Somavaratan (N=104) | rhGH (N=32)
Upper respiratory tract infection (Infections and infestations) | 12 | 3
Nasopharyngitis (Infections and infestations) | 7 | 2
Otitis media (Infections and infestations) | 7 | 0
Ear infection (Infections and infestations) | 6 | 0
Pyrexia (General disorders) | 18 | 4
Injection site pain (General disorders) | 18 | 3
Injection site haematoma (General disorders) | 6 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 12 | 5
Diarrhoea (Gastrointestinal disorders) | 7 | 1
Nausea (Gastrointestinal disorders) | 5 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 1
Headache (Nervous system disorders) | 16 | 4
Hypothyroidism (Endocrine disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
US Sites:

Institution shall cause Principal Investigator to submit a complete copy of the proposed publication to Sponsor at least 60 days prior to presentation or submission to any third party.

Non-US sites:

The Investigator and the Institution agree that any proposed publication relating to the research and/or Study conducted under this Agreement will be submitted to Sponsor for review at least 90 days prior to submission for publication.

Additional agreement conditions apply.

DOCUMENTS (2):
  • Study Protocol (2017-04-05): https://cdn.clinicaltrials.gov/large-docs/90/NCT02339090/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/90/NCT02339090/SAP_001.pdf